CLINICAL TRIAL: NCT01938001
Title: A Phase 3, Double-blind, Randomized Study to Compare the Efficacy and Safety of Rituximab Plus Lenalidomide (CC-5013) Versus Rituximab Plus Placebo in Subjects With Relapsed/Refractory Indolent Lymphoma
Brief Title: Rituximab Plus Lenalidomide for Patients With Relapsed / Refractory Indolent Non-Hodgkin's Lymphoma (Follicular Lymphoma and Marginal Zone Lymphoma)
Acronym: AUGMENT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-5013-NHL-007
Record Dates: First submitted 2013-09-05; First posted 2013-09-10 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-01

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Non-Hodgkins Follicular lymphoma, Non-Hodgkins Marginal zone lymphoma, treatment for follicular lymphoma, treatment for Marginal zone lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Rituximab; Lenalidomide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rituximab and Lenalidomide (Experimental): Participants received rituximab 375 mg/m^2 intravenously (IV) every week in Cycle 1 (Days 1, 8, 15 and 22) and on Day 1 of every 28-day cycle from Cycles 2 to 5 plus lenalidomide 20 mg by mouth (PO) once daily on Days 1 to 21 every 28 days, up to 12 cycles (21-day treatment and 7-day rest period); if creatinine clearance (CrCl) was ≥ 30 mL/min but < 60 mL/min, participants received lenalidomide 10 mg capsules on days 1 to 21 every 28 days.
  Interventions: Drug: Rituximab; Drug: Lenalidomide
- Rituximab and Placebo (Active Comparator): Participants received riituximab 375 mg/m^2 IV every week in Cycle 1 (Days 1, 8, 15 and 22) and on Day 1 of every 28-day cycle from cycle 2 to 5 plus placebo (identically matched capsule) once daily on Days 1 to 21 of every 28-day cycle up, to 12 cycles.
  Interventions: Drug: Rituximab; Drug: Placebo

INTERVENTIONS:
Drug: Rituximab — Rituximab 375mg/m^2 IV every week in Cycle 1 (Days 1, 8, 15 and 22) on Day 1 of every 28 day cycle from Cycles 2 to 5
  Other Names: Rituxan
Drug: Lenalidomide — Lenalidomide 20mg by mouth (PO) daily on Days 1 to 21 every 28 days up to 12 cycles
  Other Names: CC-5013, Revlimid
  Arms: Rituximab and Lenalidomide
Drug: Placebo — Placebo (identical matched capsule) PO daily on Days 1 to 21 every 28 days
  Arms: Rituximab and Placebo

SUMMARY:
This double-blind randomized, parallel group study will evaluate the efficacy and safety of lenalidomide (Revlimid, CC-5013) in combination with rituximab (MabThera/Rituxan) in patients with relapsed or refractory follicular lymphoma or marginal zone lymphoma. Patients will be randomized to receive either lenalidomide or placebo for twelve 28-day cycles in combination with rituximab. Anticipated time on study treatment is 1 year.

DETAILED DESCRIPTION:
Indolent lymphoma is a slow growing but incurable lymphoma which includes follicular lymphoma and marginal zone lymphoma. Follicular lymphoma and marginal zone lymphoma are cancers of the B lymphocyte, a type of white blood cell. Lenalidomide is an immunomodulatory drug (a drug that affects the immune system) which alters the body's immune system and it may also interfere with the development of tiny blood vessels involved in tumor growth. Therefore, lenalidomide may reduce or prevent the growth of cancer cells. Lenalidomide has also been shown to restore the immune cells' ability to attack and kill tumor cells, an ability that may be inhibited by follicular lymphoma and other lymphomas. The combination of rituximab and lenalidomide may eliminate the cancer while restoring the immune system's ability to attack tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years at the time of signing the informed consent document.
* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures are conducted.
* Histologically confirmed marginal zone lymphoma or follicular lymphoma (grade 1, 2 or 3a; CD20+ by flow cytometry or histochemistry).
* Previously treated with at least one prior systemic chemotherapy, immunotherapy or chemoimmunotherapy and have received at least 2 previous doses of rituximab.
* Documented relapsed, refractory or progressive disease after treatment with systemic therapy and must not be rituximab-refractory.
* Investigator considers rituximab monotherapy appropriate.
* Bi-dimensionally measurable disease on cross sectional imaging by X-ray computed tomography (CT) or magnetic resonance imaging (MRI).
* Need of treatment for relapsed, progressed or refractory disease as assessed by the investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate bone marrow function.
* Willingness to follow study visit schedule, pregnancy precautions and other protocol requirements.

Exclusion Criteria:

* Histology other than follicular or marginal zone lymphoma or clinical evidence of transformation or Grade 3b follicular lymphoma.
* Subjects taking corticosteroids during the last week prior to study treatment, unless administered at a dose equivalent to < 20 mg/day prednisone or prednisolone.
* Systemic anti-lymphoma therapy within 28 days or use of antibody agents within 8 weeks use of radioimmunotherapy within 6 months.
* Known seropositive for or active viral infection with hepatitis B virus (HBV) or/and human immunodeficiency virus (HIV).
* Known hepatitis C virus (HCV) positive with chronic HCV or active viral infection with HCV hepatitis requiring anti-viral medication (at time of randomization).
* Life expectancy < 6 months.
* Known sensitivity or allergy to murine products.
* Prior history of malignancies, other than follicular or marginal zone lymphoma, unless the subject has been free of the disease for ≥ 5 years.
* Prior use of lenalidomide.
* Known allergy to thalidomide.
* Neuropathy > Grade 1.
* Presence or history of central nervous system involvement by lymphoma.
* Subjects who are at a risk for a thromboembolic event and are not willing to take prophylaxis for it.
* Uncontrolled intercurrent illness.
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent document.
* Pregnant or lactating females.
* Any condition that places the subject at unacceptable risk if he/she were to participate in the study or that confounds the ability to interpret data from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 358 (Actual)
Dates: Start 2013-11-21 (Actual); Primary Completion 2018-06-22 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (160):
- United States (35):
  - Mitchell Cancer Center, University of South Alabama, Mobile, Alabama
  - Arizona Center for Cancer Care, Glendale, Arizona
  - Southwest Cancer Care Medical Group, Escondido, California
  - Marin Oncology Associates, Greenbrae, California
  - Wilshire Oncology Medical Group, Inc, La Verne, California
  - North County Hematology Oncology (NCHO) - TRM, LLC., Oceanside, California
  - Hematology-Oncology Medical Group of Orange County, Inc., Orange, California
  - UC Davis Medical Center, Sacramento, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Wellness Hematology Oncology, West Hills, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Florida Cancer Specialists North Region Sarah Cannon Research, St. Petersburg, Florida
  - Illinois Cancer Care, P.C., Peoria, Illinois
  - LRG Healthcare Oncology Clinic, Laconia, Indiana
  - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Louisville, J.G. Brown Cancer Center, Louisville, Kentucky
  - Providence Cancer Institute, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Coborn Cancer Center at the St. Cloud Hospital, Saint Cloud, Minnesota
  - NH Oncology - Hematology, PA, Hooksett, New Hampshire
  - The Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - University of New Mexico, Albuquerque, New Mexico
  - Weill Cornell Medical College, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Oncology Hematology Care Sarah Cannon Research, Cincinnati, Ohio
  - Local Institution - 028, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - St Francis Hospital, Greenville, South Carolina
  - Spartanburg Regional Healthcare System - Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina
  - Sarah Cannon Research Inst, Nashville, Tennessee
  - Arlington Cancer Center, Arlington, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Northwest Medical Specialties PLLC, Tacoma, Washington
- Belgium (5):
  - AZ St-Jan Brugge Oostende AV, Bruges
  - Local Institution - 371, Ghent
  - UZ Gent, Ghent
  - AZ Groeninge, Kortrijk
  - CHU Mont -Godinne, Yvoir
- Brazil (10):
  - Associacao Hospitalar Moinhos de Vento Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Associacao Educudora Sao Carlos AESC Hospital Giovanni Battista HGB Hospital Mae de Deus Center, Porto Alegre, Rio Grande do Sul
  - Fundacao Pio XII - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Hospital Dr. Amaral Carvalho/ Hospital Amaral Carvalho Jaú, Jau/SP, São Paulo
  - MS INCA HC I Hospital do Cancer I, Rio de Janeiro
  - Sociedade Beneficente de Senhoras Hospital Sirio Libanes, São Paulo
  - Real e Benemerita Associacao Portuguesa de Beneficencia, São Paulo
  - Fundação Antonio Prudente - AC Camargo Câncer center, São Paulo
- China (19):
  - Peking University People's Hospital, Beijing
  - 307 Hospital of PLA, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Beijing Cancer Hospital, Beijing, PR
  - The Third Xiangya hospital of central south university, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Fujian Medical University Union Hospital, Fuzhou
  - Sun Yat-sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Local Institution - 600, Guangzhou
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou
  - Local Institution - 604, Hangzhou
  - Jiangsu Province Hospital The First Hospital affiliated with Nanjing Medical University, Nanjing
  - Cancer Hospital, Fudan University, Shanghai
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Xijing Hospital, Xi'an
- Czechia (6):
  - Interni hematoonkologicka klinika, Brno
  - Fakultni nemocnice Hradec Kralove, IV.interni hematologicka klinika, Hradec Králové
  - Fakultni Nemocnice Ostrava, Klinika hematoonkologie,, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Interni hematologicka klinika, Prague
  - Local Institution - 534, Prague
  - Vseobecna Fakultni Nemocnice v Praze, Prague
- France (7):
  - CHU d'Angers, Angers
  - Centre Hospitalier Universitaire d'Avicennes, Bobigny
  - CHRU de Brest - Hopital Morvan, Brest
  - Hopital Saint-Louis, Paris
  - CH Perpignan - Hopital Saint-Jean, Perpignan
  - CHU de Poitiers, Poitiers
  - Centre Hospitalier de Valence, Valence
- Germany (6):
  - Charite - Universitaetsmedizin Berlin Charité - Campus Benjamin Franklin, Berlin
  - Charite - Universitaetsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Krankenhaus Nordwest, Frankfurt
  - Onkologische Schwerpunktpraxis Leer - Emden, Leer
  - Kliniken Maria Hilf GmbH, Mönchengladbach
  - Klinkum der Stadt Villingen-Schwenningen GmbH, Villingen-Schwenningen
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Hadassah University Hospital, Jerusalem
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
- Italy (16):
  - Centro di Riferimento Oncologico - IRCCS, Aviano (PN)
  - U.O.C. Ematologia, Barletta
  - A.O.U. di Bologna Policlinico S.Orsola-Malpighi, Bologna
  - Azienda Ospedaliera di Rilievo Nazionale e di Alta Specializzazione Garibaldi - Nesima, Catania
  - Istituto Scientifico Romagnolo Per Lo Studio e La Cura Dei Tumori (I.R.S.T.), Meldola
  - Istituto Europeo di Oncologia - IEO, Milan
  - Ospedale Niguarda Ca Granda, Milan
  - IRCCS- Istituto Nazionale per lo Studio e la Cura dei Tumori, Fondazione "G. Pascale", Napoli
  - Az. Osp. Vincenzo Cervello, Palermo
  - Casa di Cura La Maddalena, Palermo
  - Azienda Ospedaliero-Universitaria di Parma, Parma
  - Ospedale di Ravenna, Ravenna
  - Azienda Ospedaliera Bianchi-Melacrino-Morelli, Reggio Calabria
  - Ospedale degli Infermi di Rimini, Rimini
  - Azienda Ospedaliera S. Andrea - Università La Sapienza, Roma
  - Local Institution - 340, Roma
- Japan (13):
  - Local Institution - 708, Nagasaki, Nagasaki
  - Local Institution - 709, Minato-ku, Tokyo
  - National Cancer Center Hospital, Chūōku
  - Chugoku Central Hospital, Hiroshima
  - National Cancer Center Hospital East, Kashiwa
  - Kobe City Medical Center General Hospital, Kobe
  - The Cancer Institute Hospital of Japanese Foundation For Cancer Research, Kōtoku
  - Local Institution - 700, Kōtoku
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto
  - Toranomon Hospital, Minatoku
  - The Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Nagoya Medical Center,Division of Hematology/Oncology, Nagoya
  - National University Corporation Tohoku University, Tohoku University Hospital, Sendai
- Poland (5):
  - Malopolskie Centrum Medyczne S.C., Krakow
  - Instytut Hematologii i Transfuzjologii w Warszawie, Warsaw
  - Local Institution - 514, Warsaw
  - Centrum Onkologii, Instytut im. Marii Sklodowskiej-Curie, Warsaw
  - Local Institution - 513, Warsaw
- Portugal (4):
  - Instituto Portugues de Oncologia de Lisboa, Francisco Gentil, Lisbon
  - Local Institution - 330, Lisbon
  - Instituto Portugues de Oncologia do Porto, Francisco Gentil, Porto
  - Local Institution - 331, Porto
- Hospital Auxilio Muto Centro de Cancer, San Juan, Puerto Rico
- Russia (6):
  - Krasnoyarsk Regional Clinical Hospital, Krasnoyarsk
  - Russian Academy of Medical Sciences Institution, Moscow
  - Moscow State Medical Institution Municipal Clinical Hospital n.a. S.P. Botkin, Moscow
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Federal Centre of Heart, Blood and Endocrinology of Rosmed technlologies V.A. Almazov, Saint Petersburg
  - The Ministry of Health and Social Development of the Tula region state institution Health Tula regio, Tula
- Spain (12):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Local Institution - 314, Córdoba
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Costa del Sol, Marbella
  - Local Institution - 315, Marbella
  - Hospital Morales Meseguer, Murcia
  - Local Institution - 318, Murcia
  - Hospital Universitario de Salamanca, Salamanca
  - Local Institution - 311, Salamanca
  - Hospital Universitario Virgen Del Rocio, Seville
- Turkey (Türkiye) (8):
  - Cukurova University Medical Faculty Balcali Hospital, Adana
  - Hacettepe Universitesi, Ankara
  - Pamukkale University Medical Faculty, Denizli
  - Gaziantep University, Gaziantep
  - Marmara University, Istanbul
  - Dokuz Eylul University Izmir, Izmir
  - 19 Mayis Medical Faculty - Samsun, Samsun
  - Kocaeli Derince Training and Research Hospital, Umuttepe Kocaeli
- United Kingdom (4):
  - Eastbourne District General Hospital, Eastbourne
  - Royal Liverpool University Hospital, Prescot Street, Liverpool
  - Barts Cancer Institute, Queen Mary University of London, Charterhouse Square, London
  - Southend University Hospital NHS Foundation Trust, Prittlewell Chase, Westcliff-on-Sea

REFERENCES:
- [Background] Morschhauser F, Fowler NH, Feugier P, Bouabdallah R, Tilly H, Palomba ML, Fruchart C, Libby EN, Casasnovas RO, Flinn IW, Haioun C, Maisonneuve H, Ysebaert L, Bartlett NL, Bouabdallah K, Brice P, Ribrag V, Daguindau N, Le Gouill S, Pica GM, Martin Garcia-Sancho A, Lopez-Guillermo A, Larouche JF, Ando K, Gomes da Silva M, Andre M, Zachee P, Sehn LH, Tobinai K, Cartron G, Liu D, Wang J, Xerri L, Salles GA; RELEVANCE Trial Investigators. Rituximab plus Lenalidomide in Advanced Untreated Follicular Lymphoma. N Engl J Med. 2018 Sep 6;379(10):934-947. doi: 10.1056/NEJMoa1805104. PMID 30184451
- [Result] Leonard JP, Trneny M, Izutsu K, Fowler NH, Hong X, Zhu J, Zhang H, Offner F, Scheliga A, Nowakowski GS, Pinto A, Re F, Fogliatto LM, Scheinberg P, Flinn IW, Moreira C, Cabecadas J, Liu D, Kalambakas S, Fustier P, Wu C, Gribben JG; AUGMENT Trial Investigators. AUGMENT: A Phase III Study of Lenalidomide Plus Rituximab Versus Placebo Plus Rituximab in Relapsed or Refractory Indolent Lymphoma. J Clin Oncol. 2019 May 10;37(14):1188-1199. doi: 10.1200/JCO.19.00010. Epub 2019 Mar 21. PMID 30897038
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/safety/medwatch/safetyinformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Rituximab + Lenalidomide (R^2): Participants received rituximab 375 mg/m^2 intravenously (IV) every week in Cycle 1 (Days 1, 8, 15 and 22) and on Day 1 of every 28-day cycle from Cycles 2 to 5 plus lenalidomide 20 mg by mouth (PO) once daily on Days 1 to 21 every 28 days up to 12 cycles (21-day treatment and 7-day rest period); if creatinine clearance (CrCl) was ≥ 30 mL/min but < 60 mL/min, participants received lenalidomide 10 mg capsules on days 1 to 21 every 28 days.
- Rituximab + Placebo: Participants received rituximab 375 mg/m^2 IV every week in Cycle 1 (Days 1, 8, 15 and 22) and on Day 1 of every 28-day cycle from cycle 2 to 5 plus placebo (identically matched capsule) once daily on Days 1 to 21 of every 28-day cycle up to 12 cycles.
Period: Pre-Treatment
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Started (Started=randomized) | 178 | 180
Completed (Completed=treated) | 176 | 180
Not Completed | 2 | 0
Not completed — Adverse Event unrelated to Study Drug | 1 | 0
Not completed — Death | 1 | 0
Period: Treatment
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Started (Started=treated) | 176 | 180
Completed (Completed=completed 12 cycles of treatment) | 124 | 110
Not Completed | 52 | 70
Not completed — Death | 2 | 0
Not completed — Adverse Event | 14 | 8
Not completed — Progressive Disease | 21 | 54
Not completed — Withdrawal by Subject | 13 | 7
Not completed — Other reasons | 2 | 1

BASELINE CHARACTERISTICS:
Population: The intent to treat (ITT) population was defined as all participants who were randomized into the trial, regardless of whether they received investigational product (IP) or not.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo | Total
Number analyzed (Participants) | 178 | 180 | 358
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.30 (11.227) | 61.48 (11.160) | 61.89 (11.186)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 83 | 186
  Male | 75 | 97 | 172
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 20 | 44
  Not Hispanic or Latino | 147 | 158 | 305
  Unknown or Not Reported | 7 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 118 | 115 | 233
  Other Races | 54 | 64 | 118
  Not Collected or Reported | 6 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Kaplan Meier Estimate of Progression Free Survival Assessed by the Independent Review Committee (IRC) According to the 2007 International Working Group Response Criteria (IWGRC)
Description: Progression-free survival (PFS) was defined as the time from date of randomization into the study to the first observation of documented disease progression or death due to any cause, whichever occurred first. PFS was based on the data from the IRC review using the modified 2007 International Working Group Response Criteria (IWGRC) using FDA censoring rules.
Time Frame: From randomization of study drug up to disease progression or death, which occurred first; up to the data cut-off date of 22 June 2018; overall median follow-up time for all participants was 28.30 months (range: 0.1 to 51.3 months).
Population: The ITT population was defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
months | 39.4 [22.9 to NA] — NA =Not enough events had occurred at the time of the data cut-off date | 14.1 [11.4 to 16.7]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p < 0.0001, Log Rank; Stratified by 3 factors: previous rituximab treatment, time since last antilymphoma therapy (≤ 2, > 2 years), and disease histology (FL, MZL); Hazard Ratio (HR) = 0.46, 95% CI 2-sided [0.34 to 0.62] — Hazard ratio and its confidence interval (CI) were estimated from Cox proportional hazard model adjusting for the stratification factors noted above

2. Secondary Outcome: Durable Complete Response Rate (DCCR) as Assessed by the IRC According to the 2007 IWGRC
Description: DCCR was defined as the percentage of participants with a best response of complete response (CR) that lasted no less than one year (≥ 48 weeks) during the study prior to administration of new anti-lymphoma therapy. A CR is defined as a complete disappearance of any disease-related symptoms and normalization of biochemical abnormalities.
Time Frame: From first dose of investigational product (IP) to data cut-off date of 22 June 2018; the median treatment duration was 11.19 months in the rituximab/lenalidomiade arm and 11.04 months in the rituximab/placebo arm
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 25.3 [19.1 to 32.3] | 11.1 [6.9 to 16.6]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p = 0.0006, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Kaplan-Meier Estimate of Overall Survival (OS)
Description: Overall survival was defined as the time from randomization to death from any cause. Overall survival was censored at the last date that the participant was known to be alive for participants who were alive at the time of analysis and for participants who were lost to follow-up before death was documented.
Time Frame: From date of randomization to death due to any cause (Average of 55.71 months and a maximum up to 95.2 months)
Population: The ITT population is defined as all participants who were randomized into the trial, regardless of whether they received study treatment or not.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
Months | NA [NA to NA] — insufficient number of participants with events | NA [NA to NA] — insufficient number of participants with events
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Stratified by 3 factors: previous rituximab treatment, time since last antilymphoma therapy (≤ 2, > 2 years), and disease histology (FL, MZL); Test type: Superiority; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.37 to 0.95]

4. Secondary Outcome: Percentage of Participants With an Objective Response as Assessed by the IRC According to the 2007 IWGRC
Description: Percentage of participants with an objective response is defined as having a response of at least a PR during the study without administration of new anti-lymphoma therapy. A complete response = a complete disappearance of all detectable clinical and radiographic evidence of disease, disappearance of any disease-related symptoms, and normalization of biochemical abnormalities; a partial response (PR) = 50% decrease in SPD of the 6 largest dominant nodes or nodal masses. No increase in the size of other nodes, liver, or spleen. Splenic and hepatic nodules must regress by at least 50% in the SPD.
Time Frame: From date of first dose to data cut-off date of 22 June 2018; the median treatment duration was 11.19 months in the rituximab/lenalidomide arm and 11.04 months in the rituximab/placebo arm
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 77.5 [70.7 to 83.4] | 53.3 [45.8 to 60.8]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

5. Secondary Outcome: Percentage of Participants With a Best Response of Complete Response as Assessed by the IRC According to the 2007 IWGRC
Description: Percentage of participants with a best response of at CR during the study without administration of new anti-lymphoma therapy. A CR = Complete disappearance of all detectable clinical and radiographic evidence of disease, disappearance of any disease-related symptoms, and normalization of biochemical abnormalities.
Time Frame: From date of first dose up to data cut-off date of 22 June 2018; the median treatment duration was 11.19 months in the rituximab/lenalidomide arm and 11.04 months in the rituximab/placebo arm
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 33.7 [26.8 to 41.2] | 18.3 [13.0 to 24.8]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Kaplan-Meier Estimate of Duration of Objective Response as Assessed by the IRC According to the 2007 IWGRC
Description: Duration of response (DOR) was defined as the time from initial response (at least PR) until documented progressive disease (PD) or death. Participants who had not progressed at the time of analysis were censored at the last assessment date that the participant was known to be progression free. Participants who received a new treatment without documented progression were censored at the last assessment date that the participants was known to be progression free.
Time Frame: From randomization up to data cut-off date of 22 June 2018; overall median follow-up time for all participants was 28.30 months (range: 0.1 to 51.3 months).
Population: Participants who achieved an objective response in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 138 | 96
months | 36.6 [22.9 to NA] — Not estimable as not enough events had occurred at the time of the data cut-off date | 21.7 [12.8 to 27.6]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p = 0.0015, Log Rank; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.36 to 0.79]

7. Secondary Outcome: Kaplan-Meier Estimate of Duration of Complete Response (DOCR) as Assessed by the IRC According to the 2007 IWGRC
Description: DOCR was defined as the time from initial CR until documented PD or death. Participants who had not progressed at the time of analysis were censored at the last assessment date that the participant was known to be progression free. Participants who received a new treatment without documented progression were censored at the last assessment date that the participants was known to be progression free.
Time Frame: as for outcome 6
Population: Participants who achieved a complete response in the ITT population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 60 | 33
months | NA [25.3 to NA] — Not enough events had occurred at the time of the data cut-off date | NA [13.8 to NA] — Not enough events had occurred at the time of the data cut-off date
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p = 0.2993, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.32 to 1.43]

8. Secondary Outcome: Kaplan Meier Estimate of Event Free Survival as Assessed by the IRC According to the 2007 IWGRC
Description: Event-free survival (EFS) was defined as the time from date of randomization to date of first documented progression, relapse, institution of new anti-lymphoma treatment (chemotherapy, radiotherapy or immunotherapy) or death from any cause. Responding participants and those who were lost to follow up were censored at their last tumor assessment date.
Time Frame: From date of randomization to data cut-off date of 22 June 2018; overall median follow-up time for all participants was 28.30 months (range: 0.1 to 51.3 months).
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
months | 27.6 [22.1 to NA] — Not enough events had occurred at the time of the data cut-off date | 13.9 [11.4 to 16.7]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p < 0.0001, Stratified Log-Rank Test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.38 to 0.67] — Hazard ratio and its CI were estimated from Cox proportional hazard model adjusting for the stratification factors noted above

9. Secondary Outcome: Kaplan Meier Estimate of Time to Next Anti-Lymphoma Treatment (TTNLT)
Description: Time to next anti-lymphoma treatment (TTNLT) was defined as the time from date of randomization to date of first documented administration of a new anti-lymphoma treatment (including chemotherapy, radiotherapy, radioimmunotherapy or immunotherapy). The time to the next anti-lymphoma treatment was of special interest to the study.
Time Frame: From date of randomization to date of first documented administration of a new anti-lymphoma treatment (Average of 55.71 months and a maximum up to 95.2 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 178 | 180
Months | 73.1 [43.0 to NA] — upper limit not available due to insufficient number of participants with events | 31.8 [22.2 to 39.4]
Statistical Analysis 1: Comparison: Rituximab + Lenalidomide (R^2) vs Rituximab + Placebo; Test type: Superiority; p < 0.0001, Stratified Log Rank Test; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.39 to 0.71]

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs include AEs that started or worsened between the date of the first dose and 28 days after the date of the last dose. A serious adverse event (SAE) is any: • Death; • Life-threatening event; • Any inpatient hospitalization or prolongation of existing hospitalization; • Persistent or significant disability or incapacity; • Congenital anomaly or birth defect; • Any other important medical event. The investigator determined the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide a sufficient explanation for the event. The severity of an AE was evaluated by the investigator according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) (Version 4.03) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death
Time Frame: From first dose to 28 days post last dose (Average of 55.71 months and a maximum up to 95.2 months)
Population: The safety population was defined as all participants who have received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
Number analyzed (Participants) | 176 | 180
Participants
  Any TEAE | 174 | 173
  Any TEAE Related to Lenalidomide/Placebo (LEN/PBO) | 159 | 118
  Any TEAE Related to Rituximab (RIT) | 134 | 105
  Any Serious TEAE | 45 | 25
  Any Serious TEAE Related to LEN/PBO | 23 | 8
  Any Serious TEAE Related to RIT | 13 | 4
  Any CTCAE Grade (GR) 3/4 TEAE | 121 | 58
  Any CTCAE GR 3/4 TEAE Related to LEN/PBO | 101 | 38
  Any CTCAE GR 3/4 TEAE Related to RIT | 57 | 20
  Any GR 5 TEAE | 2 | 2
  Any TEAE Leading to Dose Reduction LEN/PBO | 46 | 6
  Any TEAE Leading to Dose Interruption LEN/PBO | 113 | 47
  Any TEAE Leading to Dose Interruption RIT | 59 | 38
  Any TEAE Leading to Discontinuation of LEN/PBO | 15 | 9
  Any TEAE Leading to Discontinuation of RIT | 6 | 2

ADVERSE EVENTS:
Time Frame: Other (Not including Serious) Adverse Events (AEs) and Serious Adverse Events (SAEs) are collected from first dose to 28 days post last dose (Average of 55.71 months and a maximum up to 95.2 months). Participants were assessed for All-cause mortality from their date of randomization to study completion (Up to approximately 100 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Rituximab + Lenalidomide (R^2) | Rituximab + Placebo
All-Cause Mortality (participants affected / at risk) | 27/178 | 47/180
Serious Adverse Events (participants affected / at risk) | 45/176 | 25/180
Other Adverse Events (participants affected / at risk) | 170/176 | 158/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Lenalidomide (R^2) (N=176) | Rituximab + Placebo (N=180)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 3 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Retinal detachment (Eye disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Volvulus (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 2 | 1
Localised oedema (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 1 | 0
Infusion related hypersensitivity reaction (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Neurosyphilis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 6 | 6
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 3 | 2
Septic shock (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Seronegative arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Transitional cell cancer of the renal pelvis and ureter localised (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 2
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 0 | 1
Adnexal torsion (Reproductive system and breast disorders) | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab + Lenalidomide (R^2) (N=176) | Rituximab + Placebo (N=180)
Anaemia (Blood and lymphatic system disorders) | 28 | 8
Leukopenia (Blood and lymphatic system disorders) | 37 | 18
Lymphopenia (Blood and lymphatic system disorders) | 8 | 14
Neutropenia (Blood and lymphatic system disorders) | 103 | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 26 | 9
Abdominal pain (Gastrointestinal disorders) | 22 | 16
Abdominal pain upper (Gastrointestinal disorders) | 11 | 7
Constipation (Gastrointestinal disorders) | 46 | 25
Diarrhoea (Gastrointestinal disorders) | 55 | 42
Dyspepsia (Gastrointestinal disorders) | 16 | 5
Nausea (Gastrointestinal disorders) | 21 | 23
Stomatitis (Gastrointestinal disorders) | 9 | 7
Vomiting (Gastrointestinal disorders) | 18 | 13
Asthenia (General disorders) | 24 | 18
Chills (General disorders) | 14 | 8
Fatigue (General disorders) | 38 | 33
Influenza like illness (General disorders) | 9 | 7
Malaise (General disorders) | 13 | 10
Oedema peripheral (General disorders) | 24 | 15
Pyrexia (General disorders) | 35 | 27
Influenza (Infections and infestations) | 17 | 8
Nasopharyngitis (Infections and infestations) | 13 | 18
Pneumonia (Infections and infestations) | 14 | 7
Sinusitis (Infections and infestations) | 13 | 5
Upper respiratory tract infection (Infections and infestations) | 33 | 23
Urinary tract infection (Infections and infestations) | 12 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 24 | 24
Alanine aminotransferase increased (Investigations) | 18 | 15
Aspartate aminotransferase increased (Investigations) | 10 | 9
Blood bilirubin increased (Investigations) | 11 | 0
Lymphocyte count decreased (Investigations) | 12 | 13
Weight decreased (Investigations) | 14 | 2
White blood cell count decreased (Investigations) | 17 | 14
Decreased appetite (Metabolism and nutrition disorders) | 23 | 11
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 11
Hyperuricaemia (Metabolism and nutrition disorders) | 10 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 15 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 18
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 10 | 12
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 | 1
Dizziness (Nervous system disorders) | 15 | 9
Headache (Nervous system disorders) | 26 | 17
Insomnia (Psychiatric disorders) | 14 | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 40 | 31
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 18 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Productive cough (Respiratory, thoracic and mediastinal disorders) | 12 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 33 | 8
Rash (Skin and subcutaneous tissue disorders) | 20 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 | 4
Hypertension (Vascular disorders) | 6 | 11
Hypotension (Vascular disorders) | 9 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-12-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT01938001/Prot_001.pdf
  • Statistical Analysis Plan (2018-06-21): https://cdn.clinicaltrials.gov/large-docs/01/NCT01938001/SAP_000.pdf